CLINICAL TRIAL: NCT06194305
Title: Multimodal Profiling of Response to Pediatric Comprehensive Behavioral Intervention for Tics
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: NEUR-2023-32286
Record Dates: First submitted 2023-10-16; First posted 2024-01-08 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-07

CONDITIONS: Tourette Syndrome; Persistent Tic Disorder
MeSH Terms: conditions — Tourette Syndrome

STUDY DESIGN:
Masking Description: This study does not involve treatment randomization so participants and all study personnel will be aware that participants are receiving CBIT. An Independent Evaluator will conduct pre-, post-treatment and 3-month follow-up assessments. This IE will be masked to information related to CBIT progress (e.g., visit attendance, specific content of sessions, therapist/supervisor perspectives on patient progress, CBIT session documentation). The IE will complete the primary outcome measure (YGTSS).
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CBIT group (Experimental): Participants with chronic TICs
  Interventions: Other: CBIT

INTERVENTIONS:
Other: CBIT — Participants will receive 8 sessions delivered weekly over 10 weeks. All sessions will be video recorded. CBIT components are: 1) Psychoeducation about tics, 2) Functional interventions, 3) Competing response (CR) training, 4) Social support: supportive people (e.g., parent, teacher) , 5) Motivational enhancements, 6) Homework: is assigned each session and typically involves self-monitoring and CR practice. Participants will complete a brief daily homework tracking log in REDCap.

SUMMARY:
Tourette Syndrome and Persistent Motor/Vocal Tic Disorder affect 1-3% of youth and can be associated with impaired functioning, emotional and behavioral problems, physical pain, diminished quality of life, and peer victimization. Chronic tics are the primary symptom. Comprehensive Behavioral Intervention for Tics (CBIT) is a manualized treatment focused on tic management skills. During the core CBIT procedure, competing response training, patients learn to inhibit tics by engaging in a competing motor action. The overall objective of this study is to identify bio-behavioral predictors and correlates of response and the most potent aspects of CBIT. Participants with chronic tics will complete a manualized course of 8-session CBIT. Neural, behavioral, psychosocial, and global functioning will be assessed longitudinally to examine predictors and correlates of response. CBIT sessions will be video recorded. CBIT process will be measured with a video-based behavioral coding scheme that will be refined and validated during years 1-2 using archival CBIT videos

ELIGIBILITY:
Inclusion Criteria:

* Age 10-17 years at time of enrollment.
* Current chronic motor and/or vocal tics, defined as tics for at least 1 year without a tic-free period of more than 3 consecutive months. Tics must not be due to a medical condition or the direct physiological effects of a substance.
* At least moderate tic severity, defined as a Yale Global Tic Severity Scale total score ≥14 (≥9 for those with motor or vocal tics only).
* Full scale IQ greater than 70.
* Child participant required to have English fluency to ensure comprehension of study measures and instructions.
* To increase external validity of findings, we will include participants taking psychotropic medications that have been stable for 6 weeks and expect to remain stable for the study period. Individuals receiving non-tic related psychotherapy involving procedures that overlap with CBIT can be eligible to participate if they refrain from receiving treatment once enrolled through the post-treatment assessment. All concurrent treatments will be monitored.

Exclusion Criteria:

* Inability to undergo MRI (e.g., metal in body, claustrophobia, orthodontia) and/or EEG.
* Active suicidality Previous diagnosis of psychosis, cognitive disability, or structural brain disease that in the investigator opinion would impede participation.
* History of seizure disorder
* Active substance abuse or dependence.
* Presence of another psychiatric or medical condition requiring immediate treatment and/or for which delay of treatment to focus on tics would be clinically inappropriate. Participants will not be excluded for comorbidities that commonly occur with TS (e.g., ADHD, OCD, anxiety) provided that this criterion is met, as only 10-15% of patients with TS have no comorbidities.
* Concurrent psychotherapy focused on tics and/or involving procedures that overlap with CBIT (e.g., habit reversal therapy, exposure therapy targeting repetitive behaviors).
* Psychotropic medication changes in the past 6 weeks and/or plans to change medication during the study period through post-treatment assessment.
* ≥ 4 previous sessions of CBIT.

Ages: 10 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2024-04-25 (Actual); Primary Completion 2029-02-19 (Estimated); Study Completion 2029-02-19 (Estimated)

PRIMARY OUTCOMES:
Change in the Total Tic Score on the Yale Global Tic Severity Scale (YGTSS). | 27 weeks
  The YGTSS is a clinician-rated measure that will be scored by a study Independent Evaluator. For each participant, the severity of tics over the past 1 week will be measured using the sing a data-dYGTSS Total Tic Score, which ranges from ranges from 0-50. Outcome will be reported as change from baseline to post-treatment, change from baseline to 1-month post-treatment, and change from post-treatment to 1-month post-treatment.

SECONDARY OUTCOMES:
Change resting-state fMRI connectivity of the brain | 27 weeks
  For each participant, signal intensity (unitless measure) will be measured using fMRI during a state of rest. Signal intensity will be measured within established resting-state brain networks. Analysis will compare within- subject change in signal intensity in these networks from pre- to post treatment; these variables will be entered into multivariate prediction models to identify the relationships between signal intensities and YGTSS Total Tic Scores.
neural, behavioral, and psychosocial changes associated with change in tic severity post-CBIT | 27 weeks
  A data- driven approach will be used to model longitudinal change across multiple key indices to inform reasons for tic severity reduction while identifying therapeutic targets that could be engaged in future research.
Quality of Life: PROMIS Pediatric Profile-49 | 27 weeks
  Description: For each participant, quality of life will be measured using the PROMIS Pediatric Profile-49 questionnaire. Each item is scored from 1-5, and scores are added together to measure overall quality of life and functioning across specific domains. Scores will be PROMIS scores will be entered into linear mixed models to see which are related to baseline YGTSS and change in baseline to post-treatment YGTSS.
Components of CBIT sessions | 27 weeks
  Recordings of CBIT session videos will be reviewed to measure the specific components of CBIT that therapists use in units of time (i.e., minutes) and frequency (e.g., number of times the therapist delivers each component across sessions). Generalized linear mixed models will be used to model the association between CBIT components and change on the YGTSS.
Identify CBIT process elements that contribute to response | 27 weeks
  code CBIT session videos to capture observable therapist and patient behaviors.

CONTACTS AND LOCATIONS:
Overall Officials: Christine Conelea, PhD, LP, Principal Investigator — University of Minnesota; Deanna Greene, PhD, Principal Investigator — University of California, San Diego; Sonya Wang, MD, Principal Investigator — University of Minnesota
Locations (2):
- United States (2):
  - University of California, San Diego, California
  - University of Minnesota, Minneapolis, Minnesota